CLINICAL TRIAL: NCT00267722
Title: A Phase 2a, Open-label Study of Visilizumab in Patients With Moderate-to-Severe Inflammatory, Nonstricturing, Nonpenetrating Forms of Crohn's Disease
Brief Title: Visilizumab for Moderate to Severe Inflammatory, Nonstricturing, Nonpenetrating Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Collaborators: PDL BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 291-412
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — visilizumab

INTERVENTIONS:
Drug: Visilizumab

SUMMARY:
The purpose of the study is to evaluate an intravenous (by injection) investigational medication to treat moderate to severe inflammatory, nonstricturing, nonpenetrating Crohn's disease. The research is being conducted at up to 5 clinical research sites in the US and Europe and is open to both men and women ages 18 to 70 years old. Participants in the study will have a number of visits to a research site up to 17 months. All study-related care and medication is provided to qualified participants at no cost: this includes all visits, examinations and laboratory work.

Visilizumab is a humanized antibody (antibodies are proteins that are normally made by the immune system to help defend the body from infections and other foreign substances) that is directed against T cells. Visilizumab selectively attacks problematic T cells and, in doing so, it may prevent them from causing inflammation. Visilizumab has also been observed to have a suppressive effect on the body's immune system (system in the body that reacts to foreign or occasionally one's own proteins).

DETAILED DESCRIPTION:
PDL BioPharma, Inc. was formerly known as Protein Design Labs, Inc.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Diagnosis of moderate-to-severe inflammatory, nonstricturing, nonpenetrating Crohn's disease, defined as Crohn's Disease Activity Index greater than or equal to 250, C-reactive protein greater than or equal to upper limit of normal, and endoscopic evidence of moderate-to-severe active inflammatory disease
* Test negative for Clostridium difficile within 3 weeks
* Signed informed consent, including permission to use protected health information

Exclusion Criteria:

* History of lymphoproliferative disorder or prior malignancy within 5 years or current malignancy
* Pregnant or nursing
* HIV, Hepatitis B or Hepatitis C infection
* Presence of obstructive symptoms, confirmed by endoscopy
* Serious infections within 12 months
* Active infections that require antibiotic therapy
* Started or changed dose of sulfasalazine, 5-aminosalicylic acid; or antibiotics, probiotics, or topical therapies for Crohn's within 2 weeks
* Serious infections that required IV antibiotic therapy or hospitalization within 8 weeks
* Increase dose of corticosteroid medication within 2 weeks
* Received a live vaccine within 6 weeks
* Received any monoclonal antibodies or investigational agents within 3 months
* Received cyclosporine or tacrolimus (FK506) within 4 weeks
* Dose change or discontinuation from 6-mercaptopurine, azathioprine, or methotrexate within 4 weeks
* Significant organ dysfunction
* Likely to require surgery in the next 6 months
* History of lymphoproliferative disorder
* History of tuberculosis or mycobacteria infection or positive chest x-ray
* History of thrombophlebitis or pulmonary embolus
* History of immune deficiency or autoimmune disorders other than Crohn's
* History of subtherapeutic blood levels of anticonvulsive medications within 1 week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Clinical response, defined as a 100-point or more decrease in Crohn's Disease Activity Index, without an accompanying increase in dose of concomitant medications, additional medications, or Crohn's Disease-related surgery.

SECONDARY OUTCOMES:
Frequency of clinical remission, duration of effect, endoscopic evidence of mucosal healing, change in C-reactive protein levels, pharmacokinetics, and immunogenicity.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Inflammatory Bowel Disease Center, Los Angeles, California
  - Mount Sinai School of Medicine, New York, New York